CLINICAL TRIAL: NCT07372196
Title: Left Bundle Branch Pacing in Patients With Hypertrophic Cardiomyopathy After Myectomy
Acronym: LEFTpaceHCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02-5/2025
Record Dates: First submitted 2026-01-01; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HCM - Hypertrophic Cardiomyopathy; Sudden Cardiac Death; Left Bundle Branch Pacing; ICD; Heart Failure (HF)
Keywords: sudden cardiac death; Hypertrophic Cardiomyopathy; Left Bundle Branch Pacing; ICD; Heart failure; myectomy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Death, Sudden, Cardiac; Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Left bundle branch area pacing (LBBAP) (Experimental): Participants assigned to Group 1 will implantation of a dual-chamber cardioverter-defibrillator with left bundle branch block pacing
  Interventions: Device: ICD with left bundle branch area pacing (LBBAP)
- Group 2: Dual-chamber cardioverter-defibrillator (Active Comparator): Participants assigned to Group 2 will implantation of a dual-chamber cardioverter-defibrillator
  Interventions: Device: dual-chamber ICD

INTERVENTIONS:
Device: ICD with left bundle branch area pacing (LBBAP) — Incision in the left or right connector area parallel to the key. Vein puncture. Electrodes are passed through the introducer system. Before implantation, a safety electrode is implanted in the LBBB at the apex of the right ventricle.
  The His bundle is recorded 1-1.5 cm apically (toward the apex of the right ventricle) in the area of the interventricular septum. Pacing from this area of the QRS complex in lead V1 has a "W" morphology. Insert the electrode into the thick interventricular septum. After each ventricular extrasystole, stop inserting and measure the following parameters:
  1. Unipolar impedance. The deeper into the septum, the lower the impedance. The target impedance is at least 500 ohms.
  2. Change the activation pattern from LBBB to RBBB.
  3. Initially, an increase, then a decrease in the unipolar signal. Fix the electrode with invisible U-shaped sutures. Control programming. Layered wound closure.
  Other Names: Left bundle branch block (LBBB) pacing
  Arms: Group 1: Left bundle branch area pacing (LBBAP)
Device: dual-chamber ICD — Under local anesthesia, an incision was made parallel to the clavicle in the left junctional area. A subcutaneous bed for the pacemaker was created. Hemostasis was maintained. The communicating vein was punctured from the wound, and through a system of introducers, it was continuously fixed in the right ventricular septum under fluoroscopic control. The electrode was fixed with a U-shaped suture. The communicating vein was again punctured, and through the system of introducers, an electrode was inserted, which was firmly fixed in the right atrial appendage under fluoroscopic control. The electrode was fixed with a U-shaped suture. The electrodes are connected to the pacemaker. Layered wound suturing is performed. An aseptic dressing is applied.
  Arms: Group 2: Dual-chamber cardioverter-defibrillator

SUMMARY:
Pilot interventional randomized clinical trial to study the efficacy of left bundle branch pacing in patients with hypertrophic cardiomyopathy after myectomy for the prevention of progression of heart failure, prevent the occurrence of life-threatening rhythm disturbances and promote reverse remodeling of the LV.

The aim of the study is to evaluate the comparative efficacy and safety of implantation of a cardioverter-defibrillator with left bundle branch block pacing and a dual-chamber cardioverter-defibrillator in patients with HCM and complete left bundle branch block after myectomy at high risk of SCD.

Objectives of the study:

1. To analyze the safety of ICD implantation procedures with LBBB pacing in patients with HCM and LBBB after myectomy at high risk of SCD;
2. To develop a technique for LBBB lead implantation in patients with HCM and LBBB after myectomy;
3. To conduct a comparative analysis of QRS complex duration data based on ECG data before and after surgery, LV activation time, and pacing threshold based on postoperative programming data;
4. To conduct a comparative analysis of the functional class of CHF, NT-proBNP, the presence/absence of interventricular and intraventricular dyssynchrony, the degree of diastolic dysfunction, LVEF, and LV EDV based on echocardiography data before and 12 months after surgery;
5. Conduct a comparative analysis of QRS complex duration data based on ECG data, LV activation time, pacing threshold, the presence of recorded episodes of AF, VT, VF, antitachycardia and shock therapy according to programming data at 3, 6, and 12 months after surgery;
6. Assess quality of life before and 12 months after surgery using the KCCQ-12 questionnaire; 30 patients (15 patients in each group) will be randomly separated into 2 groups. All participants go through ICD programming at 3, 6, and 12 months after myectomy, assessment of left ventricular remodeling based on ECG and echocardiography, NT-proBNP, assessment of quality of life before surgery and 12 months after surgery.

DETAILED DESCRIPTION:
After a discussion about the possibility of participating in the study, the patient is presented with an informed consent form and all questions of interest are explained. If consent to participate in the study is obtained, the patient and the researcher fill in all the required fields of two copies of the informed consent form and sign it. If necessary, the researcher re-explains any information regarding the study. Once informed consent has been obtained, an Individual Registration Card (IRC) is completed for the patient enrolled in the study. Completion of the IRC also continues until the completion of all stages of the study.

30 patients (15 patients in each group) will be randomly separated into 2 groups: dual-chamber ICD and a dual-chamber ICD with LBB pacing.

Initial data:

* Demographic indicators: age, gender, height, weight, body mass index;
* Disease severity: SCD risk, CHF functional class, NT-proBNP, presence/absence of interventricular and intraventricular dyssynchrony, degree of diastolic dysfunction, LVEF, LVEDV;
* Comorbidities: myocardial infarction, hypertension, diabetes mellitus, atrial fibrillation, ventricular tachycardia, chronic kidney disease, liver failure, stroke.
* The quality of life questionnaire Kansas City Cardiomyopathy Questionnaire (KCCQ-12)

Intraoperative:

* QRS complex duration according to ECG;
* LV activation time;
* Pacing threshold.

Hospitalization period:

1. Complications related to the ICD implantation procedure;
2. Adequate ICD function according to ECG and programming data.

ICD Implantation with Left Bundle Branch Pacing: Incision in the left or right connector area parallel to the key. Vein puncture. Electrodes are passed through the introducer system. Before implantation, a safety electrode is implanted in the LBBB at the apex of the right ventricle.

The His bundle is recorded 1-1.5 cm apically (toward the apex of the right ventricle) in the area of the interventricular septum. Pacing from this area of the QRS complex in lead V1 has a "W" morphology. Insert the electrode into the thick interventricular septum. After each ventricular extrasystole, stop inserting and measure the following parameters:

1. Unipolar impedance. The deeper into the septum, the lower the impedance. The target impedance is at least 500 ohms.
2. Change the activation pattern from LBBB to RBBB.
3. Initially, an increase, then a decrease in the unipolar signal. Fix the electrode with invisible U-shaped sutures. Control programming. Layered wound closure.

Statistical analysis:

Comparisons of continuous outcomes will be performed using the Mann-Whitney test for non-normal variables and the Welch t-test for normal variables. Comparisons of binary outcomes will be performed using the chi-square test or Fisher's exact test.

ELIGIBILITY:
Inclusion criteria:

* Men and women aged 18 years and older;
* Patients with post-myectomy HCM who develop LBBB with a QRS complex greater than 130 ms and a high risk of SCD (HCM Risk-SCD ≥ 6%);
* Signed informed consent to participate in the study;

Exclusion criteria:

* Absence of QRS complex morphology consistent with LBBB in LBBB with a positive QRS complex less than 130 ms;
* Presence of baseline complete RBBB;
* Heart transplantation or implantation of an LVAD is planned within the next 6 months;
* Patients with intermediate or low risk of SCD;
* History of AMI less than three months prior to study inclusion;
* Acute renal and hepatic failure;
* Acute infectious diseases;
* Presence of mental illness;
* Presence of other illnesses for which life expectancy is less than one year;
* Patient refusal to participate in the study at any stage;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 48 hours
  Absence of procedural complications requiring emergency surgical intervention (major bleeding, pneumothorax, tamponade, etc.)
Efficiency | 3-6-12 month
  Technical Success of the Procedure
  1. Reduction in QRS Duration Decrease in paced QRS duration by ≥ 20 ms compared with the baseline intrinsic QRS duration during complete left bundle branch block.
     Time Frame: At the time of implantation.
  2. QRS morphology consistent with conduction system pacing: rSR', rSr', or qR pattern in lead V1.
  Time Frame: At the time of implantation.

SECONDARY OUTCOMES:
Hospitalization for heart failure, assessment of the functional class of CH, measurement of NT-proBNP, assessment of LV remodeling, antitachycardia and shock therapy, paroxysms of supraventricular tachycardia, quality of life | 3-6-12 month
  * Hospitalization for heart failure within 12 months after ICD implantation;
  * Assessment of the functional class of CHF according to the NYHA classification at 12 months;
  * Measurement of NT-proBNP at 12 months after ICD implantation;
  * Assessment of LV remodeling (presence/absence of interventricular and intraventricular dyssynchrony) at 12 months;
  * Assessment of left ventricular end-diastolic volume at 12 months;
  * Assessment of left ventricular ejection fraction at 12 months;
  * Antitachycardia and shock therapy according to ICD programming data at 12 months;
  * Registered paroxysms of supraventricular tachycardia according to ICD programming data at 12 months;
  * Assessment of quality of life using the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) at 12 months (0 to 24 = very poor to poor; 25 to 49 = poor to fair; 50 to 74 = fair to good; and 75 to 100 = good to excellent);

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin Scientific Research Center of the Ministry of Health of Russia, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No